CLINICAL TRIAL: NCT04196790
Title: Développement d'un modèle prédictif du Risque de Survenue d'évènements Thromboemboliques Veineux Chez Les Patients Atteints de Cancer Broncho-pulmonaire métastatique
Brief Title: Development of a Model to Predict the Risk of Venous Thromboembolic Events in Patients With Metastatic Bronchopulmonary Cancer
Acronym: LUCAAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: LUCAAT ( 29BRC19. 0224)
Record Dates: First submitted 2019-12-08; First posted 2019-12-12 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Metastatic Bronchopulmonary Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Venous thrombo-embolism (VTE) is a frequent and serious complication of cancer. However, predictive tools for VTE in cancer patients is lacking.

In patients with metastatic broncho-pulmonarycancer, biochemical characteristics might help to identify patients at high risk for VTE.

The aim of this study is to derive a predictive score combining clinical and biochemical variable that predict VTE in metastatic broncho-pulmonary cancer.

DETAILED DESCRIPTION:
Venous thrombo-embolism (VTE) is a frequent and serious complication of cancer. However, predictive tools for VTE in cancer patients is lacking.

In patients with metastatic broncho-pulmonarycancer, biochemical characteristics might help to identify patients at high risk for VTE, particularly in adenocarcinoma.

The aim of this study is to derive a predictive score combining clinical and biochemical variable that predict VTE in metastatic broncho-pulmonary cancer.

ELIGIBILITY:
Inclusion Criteria:

* metastatic broncho-pulmonary cancer
* age ≥18 years
* who are eligible for chemotherapy
* non opposition obtained

Exclusion Criteria:

* age <18 years
* pregnancy, breast feeding
* VTE in the past 6 months or at the time of cancer diagnosis
* surgery in the past 3 months
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 metastatic cancer patients prospectively recruited in this prospective cohort.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-12-18 (Estimated); Study Completion 2021-12-18 (Estimated)

PRIMARY OUTCOMES:
venous thromboembolism at 12 months | 12 months
  objectively diagnosed VTE based on validated diagnostic tests

SECONDARY OUTCOMES:
overall survival | one year
  overall survival
survival without progression | one year
  survival without progression
VTE at 6 months | 6 months
  VTE at 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHRU de Brest, Brest
  - CH des Pays de Morlaix, Morlaix
  - CHIC de QUIMPER, Quimper

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning two year and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.